CLINICAL TRIAL: NCT02402673
Title: Multidimensional Diagnostics and Effect of Activity Modification in Young Adolescents With Patellofemoral Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Michael Skovdal Rathleff, Post.doc, Aalborg University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N- 20140100
Record Dates: First submitted 2015-03-12; First posted 2015-03-30 (Estimated); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Patellofemoral Pain Syndrome
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Other)
  Interventions: Other: Temporary activity modification and graded exercises

INTERVENTIONS:
Other: Temporary activity modification and graded exercises

SUMMARY:
Problem: Adolescent patellofemoral pain (PFP) is a major problem worldwide and affects 7% of adolescents. Adolescents with PFP have long-lasting severe pain and low quality of life. Current treatment is ineffective for more than 60% and new treatment approaches are needed.

Solution: A novel multidimensional diagnostic approach combining imaging, physical activity level and pain sensitisation in adolescents with PFP. This approach will enable the identification of adolescents with PFP who benefits from a new treatment strategy using activity modification to reduce loading of the patellofemoral joint and graded exercises to improve loading capacity.

DETAILED DESCRIPTION:
Participants:

Adolescents will be recruited from a population-based cohort from Aalborg and Copenhagen consisting of a total of 16 public schools. This cohort will allow for recruitment of adolescents with PFP from the following categories 1) adolescents not participating in sport outside school; 2) adolescents involved in sports a minimum of 3 times per week. In addition, a randomly recruited age- and gender-matched pain-free group from the same cohort will be recruited to form a control group.

Protocol:

All adolescents will be requested to complete an online questionnaire on current pain problems. If they report having knee pain they will be telephoned. The telephone interview will collect an anamnesis and the adolescents and their parents will be invited to a clinical examination if they have anterior knee pain with an insidious onset and with duration of more than 6 weeks. If the adolescents are diagnosed with PFP they are invited to participate in the project.

Baseline measurements:

PFP will be diagnosed using eligibility criteria in line with previous clinical trials and commonly accepted criteria. All adolescents with PFP from the cohort will be examined using self-report questionnaires, clinical examination, strength of the hip and knee, MRI and pressure pain thresholds. Pressure pain thresholds will be measured around the knee, lower leg and forearm to assess local and secondary mechanical hyperalgesia and thus the sensitisation of the central nervous pain system. Additionally, cuff-algometry will be used to asses temporal summation of pain during repeated stimuli and conditioned pain modulation. The pain-free control group will be examined using the same measurements. The comparison between adolescents with PFP and the pain-free control group will be used in 1-2 descriptive studies with the main purpose of describing this young population based on self-report questionnaires, MRI-scans, strength of the hip ad knee and pain mechanisms.

Main study:

Adolescents with PFP will be asked to participate in main study which investigates the effect of early activity modification and graded exercises among adolescents with patellofemoral pain.

Using a prospective cohort design the investigators will investigate the effect of a novel treatment strategy aimed at temporary reduction in the loading of the patellofemoral joint by activity modification. After inclusion, the custody holder and the adolescent with PFP will be informed to begin a 4 week activity modification period and avoid all sports activity including school sports. This protocol will cause a temporary reduction in the loading of the patellofemoral joint. At 4 weeks they are instructed to begin a predefined training protocol involving graded exercises. The purpose of the graded exercises is to increase loading capacity of the tissue around the knee.

ELIGIBILITY:
Inclusion Criteria:

* 10-14 years of age
* insidious onset of anterior knee or retro- patellar pain of more than 6 weeks duration
* provoked by at least two of the following situations: prolonged sitting or kneeling, squatting, running, hopping or stair climbing; tenderness on palpation of the patella, pain when stepping down or double leg squatting

Exclusion Criteria:

* Concomitant injury or pain from the hip, lumbar spine or other knee structures
* previous knee surgery
* self-reported patellofemoral instability
* current use of physiotherapy for treating knee pain
* A diagnosis of other knee conditions that may present as anterior knee pain (Mb. Osgood Schlatter, iliotibial band syndrome, sinding-larsen-Johansson, patella tendinopathy or similar).

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 152 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Self-reported recovery on 7-point Likert scale | 12 weeks.

SECONDARY OUTCOMES:
Patellofemoral Osteoarthritis Outcome Score (PFOOS) | 4 and 12 weeks and 6 and 12 months.
Pressure Pain thresholds using handheld allometry and cuff-algometry | 4 and 12 weeks.
  Pressure pain thresholds will be measured around the knee, lower leg and forearm to assess local and secondary mechanical hyperalgesia and thus the sensitisation of the central nervous pain system. In addition temporal summation and conditioned pain modulation will be measured using cuff-algometry.
Activity level. | Continuously from 0 to 4 week follow-up.
  Actigraphs activity monitors will be used to collect data on physical activity level before the intervention and after the intervention.
Isometric strength of the knee and hip. | 4 and 12 weeks.
  Isometric strength in knee extension, hip extension and hip abduction will be tested using strap-mounted dynamometry.
Self-reported recovery on 7-point Likert scale | 4 weeks, and 6 and 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Per Hölmich, Dr.Med, Study Chair — Sports Orthopedic Research Center - Copenhagen, Arthroscopic Centre Amager, Copenhagen University Hospital, Amager-Hvidovre, Denmark; Thomas Graven-Nielsen, PhD, Study Chair — Center for Sensory-Motor Interaction (SMI), Department of Health Science and Technology, Faculty of Medicine, Aalborg University, Aalborg, Denmark; Kristian Thorborg, PhD, Study Chair — Sports Orthopedic Research Center - Copenhagen, Arthroscopic Centre Amager, Copenhagen University Hospital, Amager-Hvidovre, Denmark
Locations (1):
- Aalborg Universitetshospital, Aalborg, The North Denmark Region, Denmark

REFERENCES:
- [Derived] Rathleff MS, Graven-Nielsen T, Holmich P, Winiarski L, Krommes K, Holden S, Thorborg K. Activity Modification and Load Management of Adolescents With Patellofemoral Pain: A Prospective Intervention Study Including 151 Adolescents. Am J Sports Med. 2019 Jun;47(7):1629-1637. doi: 10.1177/0363546519843915. Epub 2019 May 16. PMID 31095417